CLINICAL TRIAL: NCT07121114
Title: CAPTIVATE India - A Cross-Sectional Study to Assess the Prevalence of Cardiovascular Disease (CVD) in Individuals With Type 2 Diabetes Mellitus (T2DM) in India.
Brief Title: CAPTIVATE India - A Study to Assess the Prevalence of Cardiovascular Disease (CVD) in Individuals With Type 2 Diabetes Mellitus (T2DM) in India
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8323; U1111-1310-3556 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-08-07; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: The population consists of male and female adults who have been diagnosed with type 2 diabetes mellitus (T2DM).
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
This is a cross-sectional study assessing the prevalence of Cardiovascular Disease and describing cardio-renal risk factors among individuals with Type 2 Diabetes Mellitus in India based on medical records.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals with type 2 diabetes mellitus (T2DM), aged above or equal to 18 years.
* A confirmed diagnosis of T2DM before ethical clearance at every participating institution.
* Medical records available between 01 January 2024 to 30 September 2024 ought to have the data points required for the primary and secondary objectives. Medical records must have at least 6 months (greater than or equal to 180 days) of follow-up data from the date of diagnosis.

Exclusion Criteria:

* Diagnosis of Type 1 diabetes, or maturity-onset diabetes of the young (MODY).
* Known congenital heart disease or malformation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of male and female adults who have been diagnosed with type 2 diabetes mellitus (T2DM).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Proportion of individuals with established Cardio Vascular Disease (CVD) | From start of data collection to end of data collection (approximately 3 months)
  Proportion

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com